CLINICAL TRIAL: NCT05029921
Title: A Phase 4, Single Arm, Open-Label, 52-Week, Multicenter Study to Evaluate the Safety and Efficacy of Ustekinumab (STELARA), an Anti-Interleukin-12/23 Monoclonal Antibody, in Chinese Participants With Moderately to Severely Active Crohn's Disease
Brief Title: A Study of Ustekinumab (STELARA) in Chinese Participants With Moderately to Severely Active Crohn's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR109023; CNTO1275CRD4030 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-08-30; First posted 2021-09-01 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Ustekinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ustekinumab (Experimental): Participants will receive a single dose of ustekinumab intravenously (IV) (weight-based dose approximating 6 milligrams per kilogram [mg/kg]) at Week 0. Participants with body weight less than or equal to (<=) 55 kg will receive ustekinumab IV of 260 mg, greater than (>) 55 kg and <=85 kg will receive ustekinumab IV of 390 mg, and >85 kg will receive ustekinumab IV of 520 mg at Week 0 in induction phase followed by ustekinumab 90 mg subcutaneously (SC) in maintenance phase from Week 8 to Week 52. For participants who achieve clinical response with ustekinumab induction dosing at Week 8, will continue to receive 90 mg ustekinumab SC every 12 weeks with final dose at Week 44. If these participants meet the criteria for loss of response from Week 16 to Week 40, dose can be adjusted to 90 mg every 8 weeks (q8w). Participants who are non-responders to ustekinumab at Week 8, and achieve clinical response at Week 16, will continue to receive ustekinumab 90 mg SC q8w from Week 16 to Week 48.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — Ustekinumab will be administered as an IV injection in induction phase and as a SC injection in maintenance phase.
  Other Names: STELARA

SUMMARY:
The purpose of this study is to evaluate the clinical and endoscopic efficacy and safety of ustekinumab in Chinese participants with moderately to severely active Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Have Crohn's disease (CD) or fistulizing Crohn's disease of at least 3 months duration, with colitis, ileitis, or ileocolitis, confirmed in the past by radiography, histology, and/or endoscopy
* Have moderately to severely active CD, defined as a baseline Crohn's disease activity index (CDAI) score of greater than or equal to (>=) 220 and less than or equal to (<=) 450, and either: a. Mean daily stool frequency (SF) count >3, based on the unweighted CDAI component of the number of liquid or very soft stools or b. Mean daily abdominal pain (AP) score >1, based on the unweighted CDAI component of AP
* Have endoscopic evidence of active ileocolonic CD as assessed by central endoscopy reading at the screening endoscopy, defined as a screening simple endoscopic score for crohn's disease (SES-CD) score >=6 (or >=4 for participants with isolated ileal disease), based on the presence of ulceration in at least 1 of the 5 ileocolonic segments, resulting in the following specified ulceration component scores: a. a minimum score of 1 for the component of "size of ulcers"; and b. a minimum score of 1 for the component of "ulcerated surface"
* A woman of childbearing potential must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) at screening and a negative urine pregnancy test at baseline
* Must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study

Exclusion Criteria:

* Has complications of Crohn's disease such as symptomatic strictures or stenoses, short gut syndrome, or any other manifestation that might be anticipated to require surgery, could preclude the use of the CDAI to assess response to therapy, or would possibly confound the ability to assess the effect of treatment with ustekinumab
* Has previously demonstrated lack of initial response (that is, primary nonresponders), responded initially but then lost response with continued therapy (that is, secondary nonresponders) to Vedolizumab
* Has a history of, or ongoing, chronic or recurrent infectious disease, including but not limited to, chronic renal infection, chronic chest infection (example, bronchiectasis), recurrent urinary tract infection (example, recurrent pyelonephritis or chronic non-remitting cystitis), or open, draining, or infected skin wounds or ulcers
* History of lymphoproliferative disease, including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy or splenomegaly or monoclonal gammopathy of undetermined significance
* Has a history of severe, progressive, or uncontrolled renal, genitourinary, hepatic, hematologic, endocrine, cardiac, vascular, pulmonary, rheumatologic, neurologic, psychiatric, or metabolic disturbances, or signs and symptoms thereof

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2025-05-18 (Actual); Study Completion 2025-05-18 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Clinical Remission at Week 8 (Co-primary Endpoint) | Week 8
  Clinical remission is defined as a crohn's disease activity index (CDAI) score of less than (<) 150 (in general, CDAI score ranges from 0 to approximately 600; higher score indicates higher disease activities). CDAI will be assessed by collecting information on 8 different Crohn's disease-related variables: extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid or very soft stools, abdominal pain [AP]/cramping, use of antidiarrheal drug(s) and/or opiates, and general well-being. The last 4 variables are scored over 7 days by the participant on a diary card that participants are to complete on a daily basis.
Percentage of Participants with Endoscopic Response at Week 16 (Co-primary Endpoint) | Week 16
  Endoscopic response is defined as at least 50 percent (%) improvement from baseline in Simple Endoscopic Score for Crohn's Disease (SES-CD) score or SES-CD score less than or equal to (<=) 2. The SES-CD score is based on the evaluation of 4 endoscopic components (presence/size of ulcers, percentage of mucosal surface covered by ulcers, the percentage of affected surface, and presence/type of narrowing/strictures) across 5 ileocolonic segments. Each endoscopic component is scored from 0 to 3 for each segment, and a total score is derived from the sum of all the component scores (range, 0 [remission] to 56 [the most severe endoscopic activity]).

SECONDARY OUTCOMES:
Percentage of Participants with Clinical Remission at Week 52 (Major Secondary Endpoint) | Week 52
  Percentage of participants with clinical remission at Week 52 will be reported.
Percentage of Participants with Patient-reported Outcome (PRO)-2 Remission at Week 8 (Major Secondary Endpoint: Co-endpoint) | Week 8
  PRO-2 remission is defined as an AP mean daily score at or below 1 (AP<=1) and a stool frequency (SF) mean daily score at or below 3 (SF<=3), and no worsening of AP or SF from baseline.
Percentage of Participants with Endoscopic Remission at Week 16 (Major Secondary Endpoint: Co-endpoint) | Week 16
  Endoscopic remission is defined as SES-CD score of <= 2. The SES-CD score is based on the evaluation of 4 endoscopic components (presence/size of ulcers, percentage of mucosal surface covered by ulcers, the percentage of affected surface, and presence/type of narrowing/strictures) across 5 ileocolonic segments. Each endoscopic component is scored from 0 to 3 for each segment, and a total score is derived from the sum of all the component scores (range, 0 [remission] to 56 [the most severe endoscopic activity]).
Percentage of Participants with Endoscopic Response at Week 52 | Week 52
  Percentage of participants with endoscopic response at Week 52 will be reported.
Percentage of Participants with Endoscopic Remission at Week 52 | Week 52
  Percentage of participants with endoscopic remission at Week 52 will be reported.
Percentage of Participants with Clinical Remission at Week 3 | Week 3
  Percentage of participants with clinical remission at Week 3 will be reported.
Percentage of Participants with PRO-2 Remission at Weeks 3 and 52 | Weeks 3 and 52
  Percentage of participants with PRO-2 remission at Weeks 3 and 52 will be reported.
Percentage of Participants with Clinical Response at Weeks 3, 8, and 52 | Weeks 3, 8, and 52
  Clinical response is defined as a CDAI score decrease greater than or equal to (>=) 100 from baseline. Participants with a baseline CDAI score of >=220 to <=248 points are considered to be in clinical response if a CDAI score of <150 is attained.
Percentage of Participants with Clinical Remission at Week 52 (in Participants Induced into Clinical Remission with Ustekinumab at Week 8) | Week 52
  Percentage of participants with clinical remission at Week 52 (in participants induced into clinical remission with ustekinumab at Week 8) will be reported.
Percentage of Participants with Corticosteroid-free Remission at Week 52 | Week 52
  Corticosteroid-free remission is defined as a CDAI score <150 and not taking any corticosteroids for at least 30 days or 90 days prior to Week 52.
Change from Baseline in C-reactive Protein (CRP) Concentration at Week 3, Week 8, and Week 52 | Baseline, Week 3, Week 8, and Week 52
  Change from baseline in CRP concentration at Week 3, Week 8, and Week 52 will be reported.
Percentage of Participants with Normalization of CRP at Weeks 3, 8, and 52 | Weeks 3, 8, and 52
  Percentage of participants with normalization of CRP at Weeks 3, 8, and 52 with elevated CRP (>3.0 milligrams per liter [mg/L]) at baseline will be reported.
Change from Baseline in Fecal Calprotectin Concentration at Week 8 and Week 52 | Baseline, Week 8, and Week 52
  Change from baseline in fecal calprotectin concentration at Week 8 and Week 52 will reported. Fecal Calprotectin will be monitored as an inflammatory biomarker measured by assay.
Percentage of Participants with Normalization of Fecal Calprotectin at Weeks 8 and 52 | Weeks 8 and 52
  Percentage of participants with normalization of fecal calprotectin at Weeks 8 and 52 with elevated fecal calprotectin (>250 milligrams per kilograms [mg/kg]) at baseline will be reported.
Percentage of Participants with Fistula Response at Weeks 8 and 52 | Weeks 8 and 52
  Fistula response is defined as a >=50% reduction in the number of draining fistulas, among participants with 1 or more fistulas at baseline.
Percentage of Participants with Clinical Remission of Delayed Responders at Week 52 | Week 52
  Percentage of participants with clinical remission of delayed responders at Week 52 will be reported. Delayed responders are participants who are not in clinical response to ustekinumab at Week 8 and achieve clinical response at Week 16.
Percentage of Participants with PRO-2 Remission of Delayed Responders at Week 52 | Week 52
  Percentage of participants with PRO-2 remission of delayed responders at Week 52 will be reported.
Percentage of Participants with Clinical Response of Delayed Responders at Week 52 | Week 52
  Percentage of participants with clinical response of delayed responders at Week 52 will be reported.
Percentage of Participants with Endoscopic Response of Delayed Responders at Week 52 | Week 52
  Percentage of participants with endoscopic response of delayed responders at Week 52 will be reported.
Percentage of Participants with Endoscopic Remission of Delayed Responders at Week 52 | Week 52
  Percentage of participants with endoscopic remission of delayed responders at Week 52 will be reported.
Change from Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) Score at Week 8 and Week 52 | Baseline, Week 8 and Week 52
  IBDQ is a validated, 32-item, self-reported questionnaire for participants with IBD to evaluate PROs across 4 dimensions: bowel symptoms (loose stools, AP), systemic symptoms (fatigue, altered sleep pattern), social function (work attendance, need to cancel social events), and emotional function (anger, depression, irritability). Scores range from 32 to 224, with higher scores indicating better outcomes.
Percentage of Participants with IBDQ Response at Weeks 8 and 52 | Weeks 8 and 52
  Percentage of participants with IBDQ response (>=16-point improvement from baseline) at Weeks 8 and 52 will be reported.
Percentage of Participants with IBDQ Remission at Weeks 8 and 52 | Weeks 8 and 52
  Percentage of participants with IBDQ remission (>170-point) at Weeks 8 and 52 will be reported.
Percentage of Participants Having any Crohn's Disease (CD)-related Emergency Room (ER)/Hospitalizations (Including Surgeries) Through Week 8 and Week 52 | Weeks 8 and 52
  Percentage of participants having any CD-related ER/hospitalizations (including surgeries) through Week 8 and Week 52 will be reported.
Percentage of Participants Having any CD-related Surgery and Procedure Through Week 8 and Week 52 | Weeks 8 and 52
  Percentage of participants having any CD-related surgery and procedure through Week 8 and Week 52 will be reported.
Change from Baseline in Each of 4 Impairments from Work Productivity and Activity Impairment Questionnaire in Crohn's Disease (WPAI-CD) at Week 8 and Week 52 | Baseline, Week 8, and Week 52
  The WPAI-CD is a validated instrument created as a patient-reported quantitative assessment of the amount of absenteeism, presenteeism, and daily activity impairment attributable to CD. The WPAI-CD consists of 6 questions to determine employment status, hours missed from work due to Crohn's disease, hours missed from work for other reasons, hours worked, the degree to which Crohn's disease affected work productivity while at work, and the degree to which Crohn's disease affected activities outside of work. Four scores are derived: percentage of absenteeism, percentage of presenteeism (reduced productivity while at work), an overall work impairment score that combines absenteeism and presenteeism, and percentage of impairment in activities performed outside of work. Each of the four scores ranges from 0 to 100, with higher scores indicate greater impairment.
Percentage of Participants with a 7-point Change from Baseline in Each of 4 Impairments from WPAI-CD at Week 8 and Week 52 | Baseline, Week 8, and Week 52
  The WPAI-CD is a validated instrument created as a patient-reported quantitative assessment of the amount of absenteeism, presenteeism, and daily activity impairment attributable to CD. The WPAI-CD consists of 6 questions to determine employment status, hours missed from work due to Crohn's disease, hours missed from work for other reasons, hours worked, the degree to which Crohn's disease affected work productivity while at work, and the degree to which Crohn's disease affected activities outside of work. Four scores are derived: percentage of absenteeism, percentage of presenteeism (reduced productivity while at work), an overall work impairment score that combines absenteeism and presenteeism, and percentage of impairment in activities performed outside of work. Each of the four scores ranges from 0 to 100, with higher scores indicate greater impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (29):
- China (29):
  - Peking University Third Hospital, Beijing
  - The Military General Hospital of Beijing PLA, Beijing
  - The second Xiangya Hospital of Central South University, Changsha
  - Changzhou No 2 Peoples Hospital, Changzhou
  - West China Hospital Sichuan University, Chengdu
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - The First Affiliated Hospital Sun Yat sen University, Guangzhou
  - Guangzhou First Municipal People's Hospital, Guangzhou
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - The Second Affiliated Hospital of Zhejiang University, Hangzhou
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - Anhui Province Hospital, Hefei
  - Huzhou central hospital, Huzhou
  - Jinhua municipal central hospital, Jinhua
  - The First Affiliated Hospital of NanChang University, Nanchang
  - Zhongda Hospital Southeast University, Nanjing
  - Jiangsu Province Hospital, Nanjing
  - Ningbo medical center lihuili hospital, Ningbo
  - Huashan Hospital Fudan University, Shanghai
  - Shanghai 10th Peoples Hospital, Shanghai
  - Shanghai East Hospital, Shanghai
  - Shengjing Hospital Of China Medical University, Shenyang
  - Peking University Shenzhen Hospital, Shenzhen
  - The Second Hospital Affiliated To Suzhou University, Suzhou
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - Wuxi People s Hospital, Wuxi
  - Yangzhou First People's Hospital, Yangzhou
  - Affiliated Hospital of Zunyi Medical University, Zunyi

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency